CLINICAL TRIAL: NCT01743703
Title: Utility of Whole-body MRI (STIR and Diffusion Weighted) in the Detection of Traumatic Injuries of Undetermined Origin in Children
Brief Title: Utility of Whole-body MRI in the Detection of Traumatic Injuries of Undetermined Origin in Children
Acronym: PEDIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00393-38
Record Dates: First submitted 2011-11-04; First posted 2012-12-06 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Traumatic Injuries
Keywords: traumatic injuries; Whole-body MRI; Skeletal survey; Children; Diagnostic
MeSH Terms: conditions — Wounds and Injuries; Disease

ARMS (1):
- whole body MRI (Other): diagnostic whole body MRI, and skeletal imaging following guidelines (whole body radiographic and scintigraphic screening)
  Interventions: Other: diagnostic whole body MRI

INTERVENTIONS:
Other: diagnostic whole body MRI — diagnostic whole body MRI, both STIR and diffusion weighted

SUMMARY:
The diagnosis of abuse in children relies heavily on the presence of skeletal and extraskeletal injuries. However, some lesions are not seen by initial skeletal survey. And the investigators have to complete the skeletal survey with either bone-scan or CT scan or whole-body MRI. whole-body MRI has proved its worth in the pediatric population for the evaluation of skeletal and extraskeletal lesions in children with cancer or infectious diseases. Thus, whole-body MRI would allowed to have total picture of children without ionising radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* Infant hospitalised for sub-dural hematoma or skeletal injuries due to non accidental traumatism or skin lesions or abdominal injuries of undetermined origin

Exclusion Criteria:

* Sub-dural hematoma of accidental origin or skeletal injuries of accidental
* Origin or known origin of lesions.
* Subject already included in the study

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2016-02-13 (Actual)

PRIMARY OUTCOMES:
sensibility of MRI for detecting skeletal injuries | one week
  standard skeletal imaging is used as reference
positive predictive value of MRI for detecting skeletal injuries | one week
  standard skeletal imaging is used as reference

SECONDARY OUTCOMES:
sensibility of MRI for detecting children with skeletal injuries | one week
  standard skeletal imaging is used as reference
specificity of MRI for detecting children with skeletal injuries | one week
  standard skeletal imaging is used as reference
predictive positive value of MRI for detecting children with skeletal injuries | one week
  standard skeletal imaging is used as reference
predictive negative value of MRI for detecting children with skeletal injuries | one week
  standard skeletal imaging is used as reference

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Treguier, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France

REFERENCES:
- [Result] Proisy M, Vivier PH, Morel B, Bruneau B, Sembely-Taveau C, Vacheresse S, Devillers A, Lecloirec J, Bodet-Milin C, Dubois M, Hamonic S, Bajeux E, Ganivet A, Adamsbaum C, Treguier C; PEDIMA study research group. Whole-body MR imaging in suspected physical child abuse: comparison with skeletal survey and bone scintigraphy findings from the PEDIMA prospective multicentre study. Eur Radiol. 2021 Nov;31(11):8069-8080. doi: 10.1007/s00330-021-07896-9. Epub 2021 Apr 29. PMID 33912993